CLINICAL TRIAL: NCT05771233
Title: Effectiveness of Core Muscle Strengthening and Lumbo-pelvic Stabilization in Preventing Dance Injuries: a Randomized Clinical Trial
Brief Title: Effectiveness of Abdominal Muscle Strengthening and Pelvic Control in the Prevention of Dance Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, CRISTINA TORRES PEREZ, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 4240/2022
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Hyperlordosis; Athletic Injuries
Keywords: Dance; Arabesque; Strengthening; Lumbo-pelvic.; Core muscles; Stabilization
MeSH Terms: conditions — Swayback; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: The study design employed is a randomized clinical trial (RCT), analytical, longitudinal and prospective, with a 4 months follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention (Experimental): The group will consist of 20 participants (6 classical dancers, 4 Spanish dancers, 5 flamenco dancers and 5 contemporary dancers) who will be divided into groups according to their specialties, with a one-hour session per week for 7 weeks of physical exercise to strengthen core muscles and lumbo-pelvic stability.
  Interventions: Other: Prevention
- Control (No Intervention): The experimental group will consist of 20 participants (4 classical dancers, 6 Spanish dancers, 5 flamenco dancers and 5 contemporary dancers) who will not receive any strength training. They will be evaluated at the beginning and at the end of the study to compare the physical conditions of the participants of this group with those of the experimental group.

INTERVENTIONS:
Other: Prevention — First, an anamnesis is performed to collect information on illnesses, previous and current injuries, medication, sports practice outside of dance, diet, sleep hours and, where appropriate, information on menstruation.
  Subsequently, an individual pre-intervention assessment of each participant is carried out, where personal data is collected, motor, elasticity and flexibility, muscle strength and stability tests are performed.
  After the initial assessment, group sessions are stablished, divided by classes according to the type of specialty of 6th grade dance. The first session is focused on teaching the different exercises and the importance of muscle strengthening, the subsequent sessions are focused on the correction of the exercises, the resolution of doubts and the incorporation of progressions regarding strength and stabilization.
  At the end of the intervention, each participant is re-evaluated and results are compared.
  Arms: Prevention

SUMMARY:
Introduction. After observing the lack of lumbo-pelvic control and the difficulty in identifying the musculature used when performing the different dance positions, it was decided to carry out an exercise intervention to strengthen the abdominal musculature and lumbo-pelvic stabilization with dancers of the Dance Conservatory of Murcia. Approximately 40 students in the 6th year of professional dance of the 4 specialties taught will participate in this study.

Objectives. To improve abdominal musculature, lumbo-pelvic stability, dance technique and proprioception, to favor the correct integration of the dancer's body scheme and muscular synergies, to reduce the risk of injury and to avoid muscular compensations in the specific Arabesque dance position.

Methods. In order to develop the study, two individual and specific assessments of the dancer will be performed, pre and post intervention. In these, data and personal history were collected, assessing joint ranges and asymmetries in the movement of upper and lower limbs, and musculoskeletal assessment of the spine, hip and knee was performed by orthopedic tests. Flexibility of the ischiosural muscles will be evaluated by means of the toes-floor test and the popliteal angle test, and muscle strength in the abdominal and lumbar region for the muscles most involved in the Arabesque movement. In addition, core stability will be assessed by specific tests and hip and knee extension range along with the increase in lumbar curve when performing Arabesque.

The intervention will be carried out through group sessions of 4 to 6 participants, and exercises aimed at muscle strengthening and improving lumbo-pelvic stability will be taught. The intervention will be performed 1 hour per week, with each group, for 2 months and they will be instructed to work this routine two hours per week at home.

DETAILED DESCRIPTION:
Introduction. After observing the inefficient pelvic control and the difficulty in identifying the musculature used when performing the different dance positions, it was decided to carry out a core strengthening and lumbo-pelvic stabilization exercise intervention with dancers of the Dance Conservatory of Murcia. Approximately 40 students in the 6th year of professional dance of the 4 specialties taught will participate in this study.

Objectives. To improve core musculature, lumbo-pelvic stability, dance technique and proprioception, to favor the correct integration of the dancer's body scheme and muscular synergies, to reduce the risk of injury and to avoid muscular compensations in the specific Arabesque dance position.

Methods.For the development of the study, two individual and specific evaluations of the dancer will be performed, pre and post intervention. In them, data and personal history will be collected, assessing joint ranges and asymmetries in the movement of upper and lower limbs, and a musculoskeletal assessment of the spine, hip and knee will be performed by orthopedic tests. Flexibility of the ischiosural muscles will be evaluated by means of the toes-floor test and the popliteal angle test, and muscle strength in the abdominal and lumbar region of the muscles most involved in the arabesque movement. In addition, core stability will be evaluated by specific tests and hip and knee extension range along with hyperlordosis when performing the Arabesque.

The intervention will be carried out through group sessions of 4 to 6 participants, and exercises aimed at muscle strengthening and improving lumbo-pelvic stability will be taught. The intervention will be performed 1 hour per week, with each group, for 2 months and they will be instructed to work this routine two hours per week at home.

ELIGIBILITY:
Inclusion Criteria:

* Students in the 6th year of the Professional Dance Conservatory of Murcia.
* Dancers in the discipline of classical, contemporary, Spanish or flamenco dance.
* To have taken the subject 'Anatomy applied to Dance'.
* Sign the informed consent form.

Exclusion Criteria:

* Have any injury that currently prevents dancing.
* Have undergone surgery within the last year.
* Not attending the center regularly.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-09 (Estimated); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
muscle strength | 5 minutes.
  Is evaluated by means of the Kendall Scale, assigning a score from 0 (no muscle contraction capacity) to 5 (greater muscle contraction capacity) according to the degree of contraction and strength of the muscle evaluated. The muscles assessed have great relevance on the pelvis and favor stability when performing the Arabesque movement and other common techniques: latissimus dorsi, hip flexors (psoas major, iliacus, psoas-iliacus and psoas minor), gluteus maximus, gluteus medius, adductors, hip internal rotation (IR), hip external rotation (ER), hamstrings (distinguishing between semitendinosus and semimembranosus with respect to biceps femoris) and quadratus lumborum.
Lumbo-pelvic stability | 2 minutes.
  For use, the Star Excursion Balance Test evaluates the patient's lumbo-pelvic stability while standing on one foot.
Abdominal strength | 5 minutes.
  To assess the strength of the transversus abdominis muscle, an instrument known as Stabilizer is used to determine the pressure variation, since it starts from a pressure of 70mmHg; this instrument is used for the Prone test.
Lumbar Lordosis | One minute.
  During the performance of Arabesque, dancers tend to increase lumbar lordosis by increasing the degree of pelvic anteversion to obtain a greater degree of hip extension. This is measured in degrees with the inclinometer while the dancer executes the step.
Muscle stability | 3 minutes.
  One-leg Squat Test and Air Plane Test assess whether the subjects are able to perform a movement without losing stability. In addition, they take into account whether there is muscular compensation when performing the movement.
Stability of the lower limb. | One minute.
  The Mini Rise Test assesses whether there is a movement of the calcaneus into varus when placed in a plié position. This determines the stability of the lower limb.
Abdominal Stability. | 5 minutes.
  The Sahrmann test allows the assessment of abdominal stability when using the stabilizer. This test consists of 5 levels, with level 1 being the least stable and level 5 the most stable. The subject must perform each level until a change of pressure in the stabilizer is observed, which indicates that the individual has lost abdominal stability when performing the activity.

SECONDARY OUTCOMES:
flexibility | One minute
  is assessed by means of the toe-plant distance test, obtaining a valuation in centimeters.
visual postural analysis | 5 minutes
  static postural analysis in the three planes (frontal, coronal and transverse) to identify the presence of musculoskeletal alterations.
dynamic postural assessment | 10 minutes
  using the goniometer, a dynamic assessment is performed (degree of anterior flexion, extension, inclination and rotation), to determine if there is any postural asymmetry or movement asymmetry. Among these tests, the Adams test and the anterior flexion test are also used. At the lower limbs (MMII) level, the degree of external rotation in the in-dehors position was assessed goniometrically.
assessment of diaphragm movement | 2 minutes
  the respiratory pattern of the subjects (costal or abdomino-diaphragmatic), the existence of tension in the transversus abdominis muscle and the abdominal competence test are evaluated.
flexibility | 2 minutes
  is evaluated by means of the popliteal angle test, quantifying the measurement and classifying it according to whether it is within the normal range (<20º), grade I (20-30º) or grade II (>30º)..

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Torres Pérez, Principal Investigator — Universidad de Murcia
Locations (1):
- Professional Dance Conservatory of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith TO, Davies L, de Medici A, Hakim A, Haddad F, Macgregor A. Prevalence and profile of musculoskeletal injuries in ballet dancers: A systematic review and meta-analysis. Phys Ther Sport. 2016 May;19:50-6. doi: 10.1016/j.ptsp.2015.12.007. Epub 2016 Jan 5. PMID 27080110
- [Background] Caine D, Goodwin BJ, Caine CG, Bergeron G. Epidemiological Review of Injury in Pre-Professional Ballet Dancers. J Dance Med Sci. 2015 Dec;19(4):140-8. doi: 10.12678/1089-313X.19.4.140. PMID 26641701
- [Background] L Biernacki J, Stracciolini A, Fraser J, J Micheli L, Sugimoto D. Risk Factors for Lower-Extremity Injuries in Female Ballet Dancers: A Systematic Review. Clin J Sport Med. 2021 Mar 1;31(2):e64-e79. doi: 10.1097/JSM.0000000000000707. PMID 30589745
- [Background] Ambegaonkar JP, Caswell AM, Kenworthy KL, Cortes N, Caswell SV. Lumbar lordosis in female collegiate dancers and gymnasts. Med Probl Perform Art. 2014 Dec;29(4):189-92. doi: 10.21091/mppa.2014.4039. PMID 25433254
- [Background] Kruusamae H, Maasalu K, Wyon M, Jurimae T, Maestu J, Mooses M, Jurimae J. Spinal posture in different DanceSport dance styles compared with track and field athletes. Medicina (Kaunas). 2015 Nov;51(5):307-11. doi: 10.1016/j.medici.2015.08.003. Epub 2015 Nov 11. PMID 26674150
- [Background] Paris-Alemany A, Torres-Palomino A, Marino L, Calvo-Lobo C, Gadea-Mateos L, La Touche R. Comparison of lumbopelvic and dynamic stability between dancers and non-dancers. Phys Ther Sport. 2018 Sep;33:33-39. doi: 10.1016/j.ptsp.2018.06.010. Epub 2018 Jul 2. PMID 29982036
- [Background] Kenny SJ, Whittaker JL, Emery CA. Risk factors for musculoskeletal injury in preprofessional dancers: a systematic review. Br J Sports Med. 2016 Aug;50(16):997-1003. doi: 10.1136/bjsports-2015-095121. Epub 2015 Nov 30. PMID 26626269
- [Background] Trentacosta N, Sugimoto D, Micheli LJ. Hip and Groin Injuries in Dancers: A Systematic Review. Sports Health. 2017 Sep/Oct;9(5):422-427. doi: 10.1177/1941738117724159. Epub 2017 Aug 7. PMID 28783444
- [Background] Steinberg N, Siev-Ner I, Peleg S, Dar G, Masharawi Y, Zeev A, Hershkovitz I. Extrinsic and intrinsic risk factors associated with injuries in young dancers aged 8-16 years. J Sports Sci. 2012;30(5):485-95. doi: 10.1080/02640414.2011.647705. Epub 2012 Jan 30. PMID 22288886
- [Background] Bowerman EA, Whatman C, Harris N, Bradshaw E. A review of the risk factors for lower extremity overuse injuries in young elite female ballet dancers. J Dance Med Sci. 2015 Jun;19(2):51-6. doi: 10.12678/1089-313X.19.2.51. PMID 26045395
- See also: PREVENTION OF THE MAIN DANCE INJURIES AND MECHANISMS OF THEIR PRODUCTION — https://www.redalyc.org/pdf/3498/349853220024.pdf
- See also: The pelvis in dance — https://idus.us.es/bitstream/11441/52144/1/revista%20lidia%203%20%2821%29.pdf